CLINICAL TRIAL: NCT03291275
Title: Survival Outcomes of Uterine Malignancies in Chinese Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: SOUM-1
Record Dates: First submitted 2017-09-20; First posted 2017-09-25 (Actual); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Endometrial Neoplasms; Survival
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Death Domain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Follow-up for death and recurrence — All patients are followed up to determine definite date of diagnosis, recurrence and death.

SUMMARY:
This study aims to determine survival outcomes (overall survival and progression-free survival) of primary uterine malignancies in China and relevant risk factors in a prospective cohort study.

ELIGIBILITY:
Inclusion Criteria:

* Primary uterine malignancies.

Exclusion Criteria:

* Metastatic malignancies to uterine corpus

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with definite diagnosis of uterine malignancies in China.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years
  Survival duration from diagnosis to death
Progression-free survival | 5 years
  Survival duration from last treatment after remission to recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, China/Beiing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li L, Ma SQ, Tan XJ, Zhong S, Wu M. Pelvic Exenteration for Recurrent and Persistent Cervical Cancer. Chin Med J (Engl). 2018 Jul 5;131(13):1541-1548. doi: 10.4103/0366-6999.235111. PMID 29941707